CLINICAL TRIAL: NCT07379645
Title: PepZinGI® Crossover Heartburn Clinical Study
Brief Title: A Clinical Trial of PepZinGI® for Acute Heartburn Relief and Sleep Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NutriScience Innovations, LLC (Industry)
Collaborators: Alethios, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NSCI01
Record Dates: First submitted 2026-01-09; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heartburn
Keywords: PepZinGI; heartburn; reflux; crossover; wearable sleep metrics
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: PepZinGI (Experimental): Participants will take PepZinGI for 1 week and consume a hurdle meal. This will be followed by a 2-week washout period.
  Interventions: Dietary Supplement: PepZinGI
- Arm 2: Placebo (Experimental): Participants will take placebo for 1 week and consume a hurdle meal. This will be followed by a 2-week washout period.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PepZinGI — 75 mg patented zinc-L-carnosine complex
  Arms: Arm 1: PepZinGI
Dietary Supplement: Placebo — <0.1 mg zinc-L-carnosine
  Arms: Arm 2: Placebo

SUMMARY:
This decentralized, randomized, double-blind, placebo-controlled, two-period crossover study will evaluate whether PepZinGI® (zinc-L-carnosine) reduces food-triggered heartburn compared with placebo. Participants (N=50) complete two 1-week treatment periods (PepZinGI® and placebo) separated by a 2-week washout, for a total of 29 days. Primary outcomes are heartburn severity and frequency measured by the NutriScience Heartburn Questionnaire; secondary outcomes include PROMIS GI Reflux-13a, time to relief, rescue medication use, wearable-derived sleep metrics, Karolinska Sleep Scale, sleep diary entries, and satisfaction. All activities are remote through Alethios; no in-person visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Self-reported food-triggered heartburn with known trigger foods
* Heartburn at least once per week
* Willing to avoid OTC/supplement heartburn treatments during study (calcium-carbonate rescue allowed but must be logged and not used during hurdle-meal day/night)
* Able to complete electronic surveys and adhere to procedures
* Access to or willingness to use a compatible wearable device

Exclusion Criteria:

* Clinician-diagnosed GERD, UC, Crohn's, or IBD
* Prescribed drugs for heartburn/digestive conditions
* Heartburn less than once per week or daily throughout the month
* More than 1 alcoholic drink/day on average during study
* Recreational drug use during study
* Known allergy to zinc, L-carnosine, or study ingredients
* Pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Heartburn frequency measured by PROMIS-Gastroesophageal Reflux 13a | Baseline, Day 8, and Day 29
  Participant will select the frequency (Never, One Day, 2-6 days, Once a day, More than once a day) of heartburn related symptoms, if any. The data will be compared to baseline and day after hurdle meals for active and placebo. A lower frequency corresponds with a better outcome.
Participant sleep quality measured by Karolinska Sleep Scale | Baseline, Day 8, and Day 29
  The validated 9-point scale will measure a participant's current level of sleepiness. The data will be compared to baseline and day after hurdle meal for active and placebo. The minimum value 1 denotes "extremely alert" whereas a 9 denotes "very sleepy". A lower score corresponds with a better outcome.
Heartburn severity measured by NutriScience Heartburn Questionnaire | Day 8 and Day 29
  Participants will rank severity of heartburn related symptoms (1: None, 2: A little bit, 3: Quite a bit, 4: A lot, 5: Extremely), if any. Participant data will be compared to PepZinGI and placebo supplementation. A lower value will correspond with a better outcome.

SECONDARY OUTCOMES:
Sleep duration measured by wearable sleep devices | Baseline through Day 29
  Participant sleep duration in total hours and minutes will be acquired from wearable devices (Garmin, Apple Watch, WHOOP). Data will be compared amongst study arms. Increased sleep duration will be considered a better outcome.
Sleep quality measured by wearable sleep devices | Baseline through Day 29
  Participant sleep quality score will be acquired from wearable devices (Garmin, Apple Watch, WHOOP) with a range from 0 to 100. Data will be compared amongst study arms. Increased sleep quality score will be considered a better outcome.
Resting heart rate measured by wearable sleep devices | Baseline through Day 29
  Participant resting heart rate in beats per minute will be acquired from wearable devices (Garmin, Apple Watch, WHOOP). Data will be compared amongst study arms. Decreased resting heart rate will be considered a better outcome.
Heart rate variability measured by wearable sleep devices | Baseline through Day 29
  Participant heart rate variability reflected as time between heartbeats in milliseconds will be acquired from wearable devices (Garmin, Apple Watch, WHOOP). Data will be compared amongst study arms. Increased heart rate variability will be considered a better outcome.
Awake/restlessness moments measured by wearable sleep devices | Baseline through Day 29
  Participant awake/restlessness measured through number of awakenings throughout total sleep duration will be acquired from wearable devices (Garmin, Apple Watch, WHOOP). Data will be compared amongst study arms. Decreased awake/restlessness will be considered a better outcome.
Participant satisfaction measured by phase completion questionnaires | Day 8 and Day 29
  Participant satisfaction and perceived effectiveness will be measured by product evaluation questions (taste, recommendation level, purchasing incentive) on a sliding scale from 1 to 10 with a higher number reflecting more positive views. Data from each question will be added to obtain a satisfaction score. Increased satisfaction scores will be considered a better outcome.

IPD SHARING:
Plan to Share IPD: No